CLINICAL TRIAL: NCT04364035
Title: A Phase IIa Randomised, Double-blind, Placebo-controlled Study of HIV-1 Vaccines MVA.HTI and ChAdOx1.HTI With TLR7 Agonist Vesatolimod (GS-9620) in Early Treated HIV-1 Infection
Brief Title: Safety, Tolerability and Immunogenicity of MVA.HTI and ChAdOx1.HTI With Vesatolimod in HIV-1 Positive Patients
Acronym: AELIX-003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aelix Therapeutics (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AELIX-003
Record Dates: First submitted 2020-03-05; First posted 2020-04-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: HIV/AIDS
Keywords: HIV infection; Therapeutic Vaccines; HTI; TLR7
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — vesatolimod

STUDY DESIGN:
Intervention Model Description: double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double Blind, Two or more parties are unaware of the interventional assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CCMM+GS-9620 (Experimental): ChAdOx1.HTI 2 doses, MVA.HTI 2 doses, GS-9620 10 doses.
  Interventions: Biological: ChAdOx1.HTI; Biological: MVA.HTI; Drug: GS-9620
- PLACEBO (Placebo Comparator): ChAdOx1.HTI placebo 2 doses, MVA.HTI placebo 2 doses, GS-9620, placebo 10 doses.
  Interventions: Biological: Placebo; Drug: Placebo Oral Tablet

INTERVENTIONS:
Biological: ChAdOx1.HTI — ChAdOx1.HTI at week 0 and week 12; Vaccine delivered as one 0. 5 mL IM injection
  Arms: CCMM+GS-9620
Biological: MVA.HTI — MVA.HTI at week 24 and week 36; Vaccine delivered as one 0. 5 mL IM injection
  Arms: CCMM+GS-9620
Drug: GS-9620 — GS-9620 at week 26,28,30,32,34,38,40,42,44 and 46 Unit-dose tablet, delivered as two 3-mg tablets
  Other Names: Vesatolimod
  Arms: CCMM+GS-9620
Biological: Placebo — Saline placebo delivered as one 0. 5 mL IM injection
  Arms: PLACEBO
Drug: Placebo Oral Tablet — Unit-dose placebo tablet delivered as two 3-mg placebo tablets
  Other Names: N/H
  Arms: PLACEBO

SUMMARY:
AELIX-003 study aims to investigate the safety, tolerability, immunogenicity and efficacy of a regimen containing AELIX Therapeutics' HTI T-cell vaccines and Gilead´s Toll-Like Receptor 7 (TLR7) agonist vesatolimod in HIV-infected individuals on antiretroviral therapy. Study that will be conducted in 57 participants who have started antiretroviral therapy during early HIV infection, enrolled at various clinical trial sites in Spain. All participants will be on antiretroviral therapy upon starting the study, with their HIV viral loads <50 copies/mL. Following exposure to the vaccine/vesatolimod, all participants, under careful monitoring, will temporarily stop their antiretroviral drugs to determine if the intervention is effective in keeping their HIV levels under control.

DETAILED DESCRIPTION:
Study will evaluate safety of the investigational drugs ChAdOx1.HTI and MVA.HTI (referenced collectively as CCMM) with vesatolimod (also known as GS-9620) in participants with early treated HIV-1 infection.

The current study will also investigate the immunogenicity of CCMM + vesatolimod treatment and the impact of CCMM + vesatolimod treatment on viral rebound and viral control following an analytical treatment interruption (ATI) in participants with early treated HIV-1 infection.

HIVACAT T cell immunogen (HTI) is a novel T cell immunogen covering the most vulnerable regions of HIV. The encoding DNA sequence that has been inserted in various vaccine vectors, including viral and non-viral vectors Administration of the HTI immunogen is implemented through a heterologous prime-boost approach that includes 2 vaccine components. The aim of the sequential administration of the therapeutic vaccines is to achieve a so-called "functional cure," in which HIV-infected participants can control viral replication in the absence of ART. In this double blind, randomised, safety and tolerability study (AELIX-003), the HTI immunogen will be administered in a prime-boost regimen consisting of vaccinations with ChAdOx1.HTI (prime) and MVA.HTI (boost).

The treatment regimen in this study will also include a toll-like receptor 7 (TLR7) agonist, GS-9620, which is supported by a recent non clinical study where sequential administration of vaccines and a TLR7 agonist (GS-986, an analogue of vesatolimod) demonstrated efficacy in simian immunodeficiency virus (SIV)-infected rhesus monkeys on ART.

HTI is currently being tested in the Phase I, double blind, placebo controlled clinical study AELIX-002 through a heterologous prime-boost vaccination employing 3 products expressing the HTI antigen, DNA.HTI and MVA.HTI and ChAdOx.HTI. The available clinical data from AELIX-002 do not suggest a risk for serious adverse events (SAEs) from the products alone, used sequentially, or from the immunogen itself.

The study will screen HIV-1 infected participants who have initiated ART within 180 days (6 months) of the estimated date of HIV-1 acquisition and who have achieved virological suppression for at least 1 year prior entering AELIX-003. Participants who provide informed consent and meet study entry criteria will be randomised into 1 of 2 parallel treatment groups. The study will be conducted in 3 periods: Period 1 will last 48 weeks during which participants will receive blinded IMPs and will continue their ART regimen; Period 2 will last up to 24 weeks during which participants will discontinue their ART regimen; and Period 3 will last 12 weeks during which participants will be monitored following the restart of their ART.

ELIGIBILITY:
Inclusion Criteria:

1. Understands the study information provided and is capable of giving written informed consent, in the opinion of the investigator or designee.
2. Has confirmed HIV-1 infection.
3. Has received ART that was initiated within 6 months of the estimated date of HIV-1 acquisition. The ART regimen is required to have included ≥3 antiretroviral drugs at the time of treatment initiation and is required to include ≥3 antiretroviral drugs at screening, but temporary use of a 2-drug ART regimen during the time between ART initiation and the screening visit is permitted
4. Has plasma HIV-1 RNA levels <50 copies/mL at the screening visit and has been virologically suppressed, defined as pVL <50 copies/mL, for at least 1 year before screening; isolated blips allowed
5. Has documented stable CD4 counts ≥450 cells/mm3 for the 6 months before screening and at the screening visit.
6. Has nadir CD4 count ≥200 cells/mm3 since human immunodeficiency virus (HIV) diagnosis; isolated lower counts at the moment of acute HIV-1 infection will be allowed only if appropriate immune recovery was followed after ART initiation
7. Is ≥18 and <61 years of age on the day of screening.
8. Is willing to comply with all study procedures, including the ATI, collection of blood samples per the protocol and adherence to the ART regimen, and is available for the planned duration of the study.
9. If heterosexually active female and of childbearing potential, must be using highly effective methods of contraception from 14 days before the first vaccination until 30 days after the end of the study (or 40 days after the last dose of vesatolimod, whichever is later); all female volunteers must be willing to undergo urine pregnancy testing at the time points specified in the schedules of events.

   * Female participants who use hormonal contraceptive as one of their birth control methods must have used the same method for at least 3 months before the first vaccination.
   * Female participants who have stopped menstruating for ≥12 months but do not have documentation of ovarian hormonal failure must have a serum follicle stimulating hormone level at screening that is within the post menopausal range as provided in the Central Laboratory Manual.
10. If heterosexually active male, must use condoms or practice sexual abstinence from the screening visit until 90 days after the end of the study (or 100 days after the last dose of vesatolimod, whichever is later). Female partners of male participants must be using highly effective methods of birth control from the screening visit until 90 days after the end of the study (or 100 days after the last dose of vesatolimod, whichever is later)

Exclusion Criteria:

1. Is pregnant or lactating at the screening visit or at any time during the study or is planning on becoming pregnant over the duration of the study.
2. If available, has genotypic data (e.g., HIV genotype data) that demonstrate the presence of clinically significant mutations that would prevent the construction of a viable ART regimen post-treatment interruption.
3. Has reported multiple periods of suboptimal adherence to ART, defined as reported episodes of at least 3 days without ART that were unrelated to participation in an ATI clinical study.
4. Has a history of past ART interruptions lasting longer than 2 weeks.
5. Has participated in another interventional clinical study within 30 days before screening.
6. Has any acquired immune deficiency syndrome-defining disease or progression of HIV related disease within 90 days of screening visit.
7. Has a history of any moderate and/or severe autoimmune disease
8. Has a history or clinical manifestations of any physical or psychiatric disorder that could impair the participant's ability to complete the study.
9. Is taking HIV protease inhibitors (including low-dose ritonavir), cobicistat-containing regimens, elvitegravir, efavirenz, etravirine, or nevirapine. Participants on prohibited ART medications will be allowed to switch to an accepted treatment between screening and baseline.
10. Is taking any other concomitant treatments non compatible with vesatolimod Participants on non-compatible medications at screening (e.g., atorvastatin, proton pump inhibitors) will be allowed to switch treatments; non compatible medications must be stopped at least 30 days prior to the first dose of vesatolimod.
11. Has received approved vaccines within 2 weeks of study entry or has had a previous immunisation with any experimental immunogens within the previous 2 years.
12. Will receive any vaccines within 4 weeks prior to, or 2 weeks after, any of the planned CCMM administrations or on a week when vesatolimod is administered.
13. Has a history of anaphylaxis or a severe adverse reaction to vaccines.
14. Has received blood products within 6 months of screening.
15. Has received treatment for cancer or lymphoproliferative disease within 1 year of screening.
16. Has received any other current or prior therapy within 30 days prior to the screening visit that, in the opinion of the investigators and/or the sponsor, would make the participant unsuitable for the study or influence the results of the study.
17. Has current or has had recent use (within last 3 months before the screening visit) of IFN or systemic corticosteroids or other immunosuppressive agents (use of inhaled steroids for pulmonary conditions or topical steroids for localised skin conditions is permitted).
18. Has abnormalities of the following laboratory tests at screening:

    Haematology
    * Haemoglobin <11 g/dL (females) or 11.5 g/dL (males)
    * Absolute neutrophil count ≤1000/mm3
    * Absolute lymphocyte count ≤600/mm3
    * Platelets ≤100,000/mm3 or ≥550,000/mm3 Clinical Chemistry
    * Creatinine >1.3 × upper limit of normal (ULN)
    * Aspartate aminotransferase >2.5 × ULN
    * Alanine aminotransferase >2.5 × ULN

    Microbiology
    * Positive hepatitis B surface antigen
    * Positive for hepatitis C antibody, unless confirmed clearance of hepatitis C virus infection (spontaneous or following treatment) determined by negative serum hepatitis C virus polymerase chain reaction
    * Positive serology indicating active syphilis requiring treatment;
19. Is unwilling to undergo an ATI as planned during the study.
20. Is not suitable for inclusion in the study based on the judgment of the investigator or sponsor.
21. Current alcohol, drug, or substance abuse or history of such abuse within the 6 months prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Proportion of participants developing solicited Grade 3 or 4 local reactions | During Period 1 (Weeks 0 to 48)
  Proportion of participants developing solicited Grade 3 or 4 local reactions in the 7-day period following administration of IMPs during Period 1
Proportion of participants developing solicited Grade 3 or 4 systemic reactions | During Period 1 (Weeks 0 to 48)
  Proportion of participants developing solicited Grade 3 or 4 systemic reactions in the 7-day period following administration of IMPs during Period 1
Proportion of participants developing treatment-emergent SAEs | During Period 1 (Weeks 0 to 48)
  Proportion of participants developing treatment-emergent SAEs during Period 1

SECONDARY OUTCOMES:
Proportion of participants who achieve virologic suppression after resumption of ART | After period 1(Week 48 to week 84)
  Proportion of participants who achieve virologic suppression (<50 copies/mL) after resumption of ART at Week 84
Proportion of participants developing treatment-emergent adverse events and SAEs (TEAEs) | After period 1(Week 48 to week 84)
  Proportion of participants developing treatment-emergent adverse events and SAEs (TEAEs)
Proportion of participants with viral load <50 copies/mL/ <2000 copies/mL at 12 and 24 weeks after the start of ATI | Week 48 to week 72
  Proportion of participants with viral load <50 copies/mL/ <2000 copies/mL at 12 and 24 weeks after the start of ATI
Proportion of participants that remain off ART at 12 and 24 weeks after the start of ATI | Week 48 to week 72
  Proportion of participants that remain off ART at 12 and 24 weeks after the start of ATI
Breadth of total vaccine-induced HIV 1-specific responses | Period1 (week 0 to 48)
  Breadth of total vaccine-induced HIV 1-specific T cell responses measured IFN-γ ELISPOT in vaccine and placebo recipients.
Proportion of participants with T cell responses to HTI encoded regions infection | Period1 (week 0 to 48)
  Proportion of participants withT cell responses to HTI encoded regions

OTHER OUTCOMES:
Evaluate the pharmacodynamic (PD) in Serum /plasma cytokines of GS-9620 | week 26- week 46
  Changes from baseline in serum/plasma cytokines.
Evaluate the pharmacodynamic (PD) in gene expression of GS-9620 | week 26- week 46
  Changes from baseline in gene expression, including ISGs (interferon stimulation genes).
Evaluate the pharmacodynamic (PD) effects of GS-9620 | week 26- week 46
  Changes from baseline in immune cell phenotype/activation in peripheral blood measured with Flow Cytometry
Maximum concentration (Cmax) of plasma GS-9620 | week 26 to week 46
  Evaluation of plasma pharmacokinetics of GS-9620 concentration data using Cmax (maximum observed concentration of drug).
Last measurable plasma concentration (Clast) of plasma GS-9620 | week 26 to week 46
  Evaluation of plasma pharmacokinetics of GS-9620 concentration data using Clast ( last observed quantifiable plasma concentration of the drug).
Time of maximum concentration (Tmax) of plasma GS-9620 | week 26 to week 46
  Evaluation of plasma pharmacokinetics of GS-9620 concentration data using Tmax: time (observed time point) of Cmax.
Terminal half-life (t1/2) of plasma GS-9620 | week 26 to week 46
  Evaluation of plasma pharmacokinetics of GS-9620 concentration data using t1/2 estimate of the terminal elimination half-life of the drug in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Arribas Lopez, Md, PhD, Study Chair — Hospital Universitario La Paz
Locations (9):
- Spain (9):
  - IrsiCaixa AIDS Research Institute, Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid